CLINICAL TRIAL: NCT03891212
Title: The Effect of Prone Position Drainage on the Efficacy of Severe Pneumonia，a Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81770081
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Severe Pneumonia
Keywords: Prone Position; Treatment Outcome; Respiration, Artificial
MeSH Terms: conditions — Pneumonia; Respiratory Aspiration | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Using a central randomization system, participants will be randomized (1:1) into groups receiving either placed in prone position or in supine position (within 24 h of diagnosis of SP) for 5-7 days with a 28-day follow-up. Patients assigned to the prone group had to be turned within the first hour following randomization. They were placed in prone position for at least 16 consecutive hours.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The prone group (Experimental): Patients assigned to the prone group had to be turned within the first hour following randomization. They were placed in prone position for at least 16 consecutive hours.
  Interventions: Behavioral: Placed in prone position for at least 16 consecutive hours a day.
- The supine group (No Intervention): Patients assigned to the supine group had to be turned within the first hour following randomization. They were placed in supine position for at least 16 consecutive hours.

INTERVENTIONS:
Behavioral: Placed in prone position for at least 16 consecutive hours a day. — Patients assigned to the prone group had to be turned within the first hour following randomization. They were placed in prone position for at least 16 consecutive hours. Patients assigned to the control group had to be turned within the first hour following randomization. They were placed in supine position for at least 16 consecutive hours.
  Arms: The prone group

SUMMARY:
Enrollment criteria and clinical data collection: follow the principles of medical ethics, the development of inclusion and exclusion criteria, Select all eligible patients with severe pneumonia(SP) who were admitted to the hospital during the study date.The diagnostic criteria we will use for SP are based on the Infectious Diseases Society of America/American Thoracic Society guidelines.Primary outcome measures：a.CURB-65 Score for Pneumonia Severity;b.The changes in inflammation and coagulation indicators: C-reactive protein, procalcitonin, and d-dimer;c.Chest x-ray changes;d.Mortality rate after 28 days;e.The time of mechanical ventilation, total duration of ICU stay, hospitalization, and antibiotic use;f.The time of bacterial cultures becoming negative;g.Daily sputum drainage.The aim of this study is to evaluate the anti-infective effectiveness and safety of prone position drainage compared with supine position on SP treatment.

DETAILED DESCRIPTION:
Severe pneumonia (SP) is a major complication of respiratory system diseases that is associated with high mortality and morbidity. If not treated correctly, it may rapidly lead to sepsis and multiple organ dysfunction syndrome. Randomized, controlled trials have confirmed that oxygenation is significantly better when patients are in the prone position than when they are in the supine position.But whether prone drainage is beneficial for rapid infection control on SP treatment has not been researched.The aim of this study is to evaluate the anti-infective effectiveness and safety of prone position drainage compared with supine position on SP treatment.

Using a central randomization system, participants will be randomized (1:1) into groups receiving either placed in prone position or in supine position (within 24 h of diagnosis of SP) for 5-7 days with a 28-day follow-up. Patients assigned to the prone group had to be turned within the first hour following randomization. They were placed in prone position for at least 16 consecutive hours.

The patients enrolled in this study should meet the diagnostic and inclusion criteria and provide written informed consent.

Diagnostic criteria The diagnostic criteria we will use for SP are based on the Infectious Diseases Society of America/American Thoracic Society guidelines.

The inclusion criteria are as follows:

1.Age ≥18 years and ≤75 years, male or female；2.Weight ≥40 kg and ≤100 kg；3.Meet the diagnostic criteria for SP；4.Need invasive mechanical ventilation；5.Provide signed informed consent

Non-inclusion criteria:

1. Contraindication for prone positioning

   a. Intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mmHg;b. Massive hemoptysis requiring an immediate surgical or interventional radiology procedure; c. Tracheal surgery or sternotomy during the previous 15 days;d. Serious facial trauma or facial surgery during the previous 15 days;e. Deep venous thrombosis treated for less than 2 days; f. Cardiac pacemaker inserted in the last 2 days;g. Unstable spine, femur, or pelvic fractures;h. Mean arterial pressure lower than 65 mm Hg;i. Pregnant women; j. Single anterior chest tube with air leaks.
2. Respiratory reason

   1. Inhaled nitric oxide (NOi) or almitrine bismesylate use before inclusion;b. Use of extracorporeal membrane oxygenation (ECMO) before inclusion.
3. Clinical context a. Lung transplantation;b. Burns on more than 20 % of the body surface;c. Chronic respiratory failure requiring oxygen therapy or non-invasive ventilation(NIV);d. Underlying disease with a life expectancy of less than one year;e. NIV delivered for more than 24 hours before inclusion.
4. Other non-inclusion criteria a. End-of-life decision before inclusion;b. Inclusion in another research protocol in the previous 30 days with mortality as the main end-point;c. Prone positioning before inclusion;d. Subject deprived of freedom, minor, subject under a legal protective measure;e. Opposition from next of kin.

Suspension criteria

The criteria for suspension of participation are as follows:

1.Poor compliance of investigators or patients;2.Occurrence of serious adverse events (AEs), complications, or fatal physiological changes;3.Voluntary withdrawal;4.Incomplete data; Primary outcome measures：

a.CURB-65 Score for Pneumonia Severity;b.The changes in inflammation and coagulation indicators: C-reactive protein, procalcitonin, and d-dimer;c.Chest x-ray changes;d.Mortality rate after 28 days;e.The time of mechanical ventilation, total duration of ICU stay, hospitalization, and antibiotic use;f.The time of bacterial cultures becoming negative;g.Daily sputum drainage.

The statistical analysis will be performed using SAS software version 9.4 (SAS Institute, Cary, NC, USA). If the lower limit of the 95 % confidence interval is larger than a clinically meaningful difference, therapeutic effects of the experimental group are deemed to be clinically and statistically better than those of the control group. Two-sided tests will be performed for all the other statistical analyses. Cochran-Mantel-Haenszel χ2 tests or Fisher's exact tests will be used for comparison of categorical outcomes. Continuous outcomes will be analyzed by using Student's t test. p values ˂0.05 are considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years, male or female
* Weight ≥40 kg and ≤100 kg
* Meet the diagnostic criteria for SP
* Need invasive mechanical ventilation
* Provide signed informed consent

Exclusion Criteria:

* Contraindication for prone positioning：a. Intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mmHg;b. Massive hemoptysis requiring an immediate surgical or interventional radiology procedure; c. Tracheal surgery or sternotomy during the previous 15 days;d. Serious facial trauma or facial surgery during the previous 15 days;e. Deep venous thrombosis treated for less than 2 days; f. Cardiac pacemaker inserted in the last 2 days;g. Unstable spine, femur, or pelvic fractures;h. Mean arterial pressure lower than 65 mm Hg;i. Pregnant women; j. Single anterior chest tube with air leaks.
* Respiratory reason：a. Inhaled nitric oxide (NOi) or almitrine bismesylate use before inclusion;b. Use of extracorporeal membrane oxygenation (ECMO) before inclusion.
* Clinical context：a. Lung transplantation;b. Burns on more than 20 % of the body surface;c. Chronic respiratory failure requiring oxygen therapy or non-invasive ventilation(NIV);d. Underlying disease with a life expectancy of less than one year;e. NIV delivered for more than 24 hours before inclusion.
* Other non-inclusion criteria ：a. End-of-life decision before inclusion;b. Inclusion in another research protocol in the previous 30 days with mortality as the main end-point;c. Prone positioning before inclusion;d. Subject deprived of freedom, minor, subject under a legal protective measure;e. Opposition from next of kin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The changes in C-reactive protein | On the tenth day after hospitalization
  Use C-reactive protein to assess the patient's lung infection status
The changes in procalcitonin | On the tenth day after hospitalization
  Use procalcitonin to assess the patient's lung infection status
The changes in d-dimer | On the tenth day after hospitalization
  Use d-dimer to assess the patient's lung infection status
Chest x-ray changes | On the tenth day after hospitalization
  Use Chest x-ray to assess the patient's lung infection status
Mortality rate after 28 days | 28 days after admission
  Calculate patient 28-day mortality
The time of total duration of ICU stay | 28 day
  Calculate The time of total duration of ICU stay
The time of mechanical ventilation | 28 day
  Calculate The time of mechanical ventilation
mortality | 28 day
  Using the Kaplan-Meier method to analyze the differences in mortality between the two groups within 28 days
The time of antibiotic use | 28 day
  Calculate the time of antibiotic use
The time of bacterial cultures becoming negative | 28 day
  Calculate the time of bacterial cultures becoming negative
Daily sputum drainage | On the tenth day after hospitalization
  Calculate daily sputum drainage

CONTACTS AND LOCATIONS:
Overall Officials: Pinhua Pan, Doctor, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China